CLINICAL TRIAL: NCT00004065
Title: A Phase I Trial of 17-N-Allylamino-17-Demethoxy Geldanamycin (17-AAG, NSC #330507) Daily X 5 in Patients With Advanced Cancer Therapeutic Protocol
Brief Title: Chemotherapy in Treating Patients With Refractory Advanced Solid Tumors or Hematologic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 99-037; CDR0000067267 (Registry Identifier: PDQ (Physician Data Query)); NCI-T99-0035; UCLA-0206019
Record Dates: First submitted 1999-12-10; First posted 2003-01-27 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Bladder Cancer; Breast Cancer; Colorectal Cancer; Gastric Cancer; Head and Neck Cancer; Kidney Cancer; Leukemia; Lung Cancer; Melanoma (Skin); Ovarian Cancer; Prostate Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage III colon cancer; stage IV colon cancer; stage IV breast cancer; stage IIIA breast cancer; recurrent breast cancer; stage III gastric cancer; stage IV gastric cancer; recurrent gastric cancer; stage IIIB breast cancer; stage IIIC breast cancer; recurrent non-small cell lung cancer; recurrent colon cancer; stage III renal cell cancer; stage IV renal cell cancer; recurrent renal cell cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; stage III bladder cancer; recurrent bladder cancer; stage IV bladder cancer; stage III prostate cancer; stage IV prostate cancer; recurrent prostate cancer; stage III melanoma; stage IV melanoma; recurrent melanoma; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; unspecified adult solid tumor, protocol specific; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; untreated metastatic squamous neck cancer with occult primary; recurrent metastatic squamous neck cancer with occult primary; ovarian stromal cancer; stage III ovarian germ cell tumor; stage IV ovarian germ cell tumor; recurrent ovarian germ cell tumor; stage III squamous cell carcinoma of the lip and oral cavity; stage III basal cell carcinoma of the lip; stage III mucoepidermoid carcinoma of the oral cavity; stage III adenoid cystic carcinoma of the oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage IV basal cell carcinoma of the lip; stage IV verrucous carcinoma of the oral cavity; stage IV mucoepidermoid carcinoma of the oral cavity; stage IV adenoid cystic carcinoma of the oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; recurrent basal cell carcinoma of the lip; recurrent verrucous carcinoma of the oral cavity; recurrent mucoepidermoid carcinoma of the oral cavity; recurrent adenoid cystic carcinoma of the oral cavity; stage III squamous cell carcinoma of the oropharynx; stage III lymphoepithelioma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; stage IV lymphoepithelioma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; recurrent lymphoepithelioma of the oropharynx; stage III squamous cell carcinoma of the nasopharynx; stage III lymphoepithelioma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; stage IV lymphoepithelioma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; recurrent lymphoepithelioma of the nasopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage III verrucous carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage IV verrucous carcinoma of the larynx; recurrent squamous cell carcinoma of the larynx; recurrent verrucous carcinoma of the larynx; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage III inverted papilloma of the paranasal sinus and nasal cavity; stage III midline lethal granuloma of the paranasal sinus and nasal cavity; stage III esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV inverted papilloma of the paranasal sinus and nasal cavity; stage IV midline lethal granuloma of the paranasal sinus and nasal cavity; stage IV esthesioneuroblastoma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent inverted papilloma of the paranasal sinus and nasal cavity; recurrent midline lethal granuloma of the paranasal sinus and nasal cavity; recurrent esthesioneuroblastoma of the paranasal sinus and nasal cavity; borderline ovarian surface epithelial-stromal tumor; ovarian sarcoma; stage III verrucous carcinoma of the oral cavity; recurrent salivary gland cancer; stage IV salivary gland cancer; stage III salivary gland cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Breast Neoplasms; Colorectal Neoplasms; Stomach Neoplasms; Head and Neck Neoplasms; Kidney Neoplasms; Leukemia; Lung Neoplasms; Melanoma; Ovarian Neoplasms; Prostatic Neoplasms; Colonic Neoplasms; Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell; Carcinoma, Ovarian Epithelial; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Squamous Cell Carcinoma of Head and Neck; Esthesioneuroblastoma, Olfactory; Salivary Gland Neoplasms | interventions — tanespimycin

INTERVENTIONS:
Drug: tanespimycin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: This phase I trial is studying the side effects and best dose of 17-N-allylamino-17-demethoxygeldanamycin in treating patients with refractory advanced solid tumors or hematologic cancers.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of 17-N-allylamino-17-demethoxygeldanamycin (17-AAG) in patients with refractory or advanced solid tumors or hematologic malignancies.
* Evaluate the effects of this drug on the expression of signaling proteins present on an individual patient's cancer at the start of treatment and, if possible, post treatment.

OUTLINE: This is a two-phase, dose-escalation, multicenter study. Patients are stratified according to disease (chronic myelogenous leukemia [CML] or Philadelphia chromosome [Ph]+ acute lymphoblastic leukemia [ALL] vs solid tumor).

Patients receive 17-N-allylamino-17-demethoxygeldanamycin (17-AAG) IV over 60-90 minutes twice weekly. Courses repeat every 12 weeks in the absence of disease progression (after at least 2 courses for CML or Ph+ ALL patients) or unacceptable toxicity.

* Accelerated phase: Single patients receive escalating dose levels of 17-AAG until one patient experiences a first course grade 3 or greater toxicity or two different patients experience grade 2 toxicity during any course.
* Standard phase: Cohorts of 3-6 patients in each stratum receive escalating doses of 17-AAG until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: Approximately 51 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following:

  * Histologically confirmed advanced primary or malignant solid tumor refractory to standard therapy or for which no curative standard therapy exists

    * Progressive disease evidenced by 1 of the following:

      * Non-prostate cancer (including, but not limited to, breast, ovary, head and neck, non-small cell lung, bladder, kidney, colon, stomach, or malignant melanoma)

        * Development of new lesions or an increase in existing lesions
        * No increase in a biochemical marker (e.g., carcinoembryonic antigen, CA-15-3, or an increase in symptoms) as sole measure of disease
  * Prostate cancer (androgen independent) meeting the following criteria:

    * Progressing metastatic disease on bone scan, CT scan, or MRI
    * Metastatic disease and rising prostate-specific antigen (PSA) values meeting 1 of the following criteria:

      * At least 3 rising PSA values obtained at least 1 week apart = 2 rising values more than 1 month apart with at least 25% increase over the range of values
    * Serum testosterone less than 30 ng/mL
    * Castrate status should be maintained by medical therapies if orchiectomy has not been performed
    * Progressive disease must be evident off antiandrogen therapy if received prior to study entry
    * Registered to protocol MSKCC-9040
  * Cytologically confirmed chronic, accelerated, or blastic phase chronic myelogenous leukemia (CML) or Philadelphia chromosome (Ph)-positive acute lymphoblastic leukemia (ALL) refractory to standard therapy or for which no curative therapy exists

    * Progressive disease evidenced by 1 of the following:

      * Accelerated or blastic phase disease that is not responsive to standard therapy or loss of hematologic response to imatinib mesylate while remaining in chronic phase for CML
      * Relapsed or refractory after treatment with standard chemotherapy and imatinib mesylate for Ph-positive ALL
* No active CNS or epidural tumor
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Not specified

Menopausal status:

* Not specified

Performance status:

* Karnofsky 70-100%

Life expectancy:

* At least 6 months

Hematopoietic:

* WBC greater than 3,500/mm^3
* Platelet count greater than 100,000/mm^3
* No restrictions based on peripheral blood counts for CML and Ph-positive ALL

Hepatic:

* Bilirubin no greater than 1.2 times upper limit of normal (ULN)
* AST less than 1.5 times ULN
* Prothrombin time normal

Renal:

* Creatinine no greater than 1.5 times ULN OR
* Creatinine clearance greater than 60 mL/min

Cardiovascular:

* No myocardial infarction within the past 6 months
* Ejection fraction greater than 45% by radionuclide cardiac angiography
* No ventricular aneurysm or other abnormal wall motion
* No reversible defect by thallium stress test if any of the following conditions are present:

  * Ejection fraction less than 45% on radionuclide angiocardiography
  * Worrisome but nonexclusive cardiovascular history
  * Abnormal echocardiogram
* Patients with the following history or clinical findings require additional diagnostic testing:

  * Significant Q waves (greater than 3 mm or greater than one-third of the height of the QRS complex)
  * ST elevation or depressions of greater than 2 mm that are not attributable to hypertension strain
  * Absence of regular sinus rhythm
  * Bundle branch block
  * Requirement for diuretics for reasons other than hypertension or digoxin for reasons other than atrial fibrillation
  * Prior mild to moderate congestive heart failure
* No New York Heart Association class III or IV heart disease
* No angina pectoris
* No uncontrolled hypertension or intermittent claudication
* No severe debilitating valvular disease

Pulmonary:

* No severe debilitating pulmonary disease

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active infection requiring IV antibiotics
* No symptomatic peripheral neuropathy grade 2 or higher
* No other severe medical conditions that would increase risk for toxicity
* No allergy to eggs or egg products

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior biologic therapy (including interferon for CML) and recovered

Chemotherapy:

* At least 4 weeks since prior chemotherapy (3 days for hydroxyurea for CML or ALL) and recovered
* No other concurrent chemotherapy

Endocrine therapy:

* See Disease Characteristics
* At least 4 weeks since prior endocrine therapy and recovered

Radiotherapy:

* At least 4 weeks since prior radiotherapy and recovered
* Concurrent radiotherapy to localized disease sites not being used to evaluate antitumor response allowed
* No concurrent radiotherapy to only measurable lesion

Surgery:

* See Disease Characteristics
* Prior orchiectomy allowed
* No concurrent surgery

Other:

* At least 3 days since prior imatinib mesylate for CML or ALL
* At least 4 weeks since prior investigational anticancer drugs and recovered
* At least 4 weeks since prior palliative treatment for metastatic disease
* No concurrent ketoconazole, warfarin, verapamil, miconazole, or erythromycin
* No other concurrent investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-07; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard I. Scher, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Memorial Sloan-Kettering Cancer Center, New York, New York